CLINICAL TRIAL: NCT04407325
Title: Tuberculosis Screening With AeoNose and CAD4TB in Paraguayan Prisons
Brief Title: Tuberculosis Screening in Paraguayan Prisons
Acronym: Prinose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: European Union (Other); Instituto de Saude Publica da Universidade do Porto (Other); VHIR (Unknown); University Medical Center Groningen (Other); Laboratorio central de salud publica, Paraguay (Unknown); Instituto Nacional de Enfermedades Respiratorias y del Ambiente Juan Max Boetner (Unknown); National TB program Paraguay (Unknown); IICS Paraguay (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 823890-EUSAT-RCS
Record Dates: First submitted 2020-04-23; First posted 2020-05-29 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Volatile Organic Compounds; Radiography
Keywords: tuberculosis; vulnerable populations; screening algorithms; cost effectiveness; neural networks; artificial intelligence
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: outcomes of individual smell prints and digital ChestXrays will be compared with sputum sampling for GenXpert and Mycobacterial culture
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AeoNose (Experimental): the AeoNose will be compared with digital ChestXray and the conventional methods of establishing TB diagnosis
  Interventions: Device: electronic nose device; Device: dig chest Xray with automated readings

INTERVENTIONS:
Device: electronic nose device — electronic nose device will be tested as a triage instrument for tuberculosis in a high risk population
  Other Names: (AeoNose, The eNose Company, the Netherlands)
Device: dig chest Xray with automated readings — software for tuberculosis detection on digital Chest Xray providing a probability score from 0-100
  Other Names: CAD4TB computed automated detection software

SUMMARY:
Two diagnostic tools for TB screening in high risk groups need additional assessment: the AeoNose™, an 'electronic nose device' for breath sampling, and digital chest X-ray (CXR) with computer aided detection with CAD4TB® software. This study will systematically screen prisoners and its' employees for TB, test the diagnostic performance of AeoNose™ and CAD4TB (both individually and together) as a TB screening tool and and establish Mycobacterium tuberculosis epidemiology in Paraguayan prisons.

DETAILED DESCRIPTION:
The aim of the World Health Organization (WHO) "End TB Strategy" is to end the global pandemic by 2035. To be able to succeed, better point-of-care (POC) tests are urgently needed to improve screening of high-risk populations. Prisons are recognized worldwide as high risk environments for the concentration, amplification and transmission of TB among prisoners and their communities outside. Paraguayan penal institutions are known to have very high incidence rates of active TB (3000-5000/100.000, according to Paraguayan Ministry of Justice). Two diagnostic tools for TB screening in high risk groups will be evaluated: the AeoNose™, an 'electronic nose device' for breath sampling, and digital chest X-ray (CXR) with computer aided detection with CAD4TB® software. This study will systematically screen prisoners and its' employees for TB, test the diagnostic performance of AeoNose™ and CAD4TB® and assess prison Mycobacterium tuberculosis epidemiology through several objectives: Objective: 1. Assessment of the sensitivity and specificity of the AeoNose™ and its utility for mass TB screening in high incidence settings. 2. Evaluation of the feasibility and utility of CAD4TB® digital CXR as a mass screening tool for TB. 3. Identification of factors that affect diagnostic accuracy of AeoNose™ and CAD4TB®. 4. Assessment of TB epidemiology in Paraguayan prisons and identification of mycobacterial strains.

Study design: Diagnostic cohort study. Study population: Detainees (PPL) of Paraguayan penal institutions as well as their employees. Nature and extent of the burden and risks associated with participation, benefit and group relatedness.

Individual burden: all participants will perform one visit with a medical doctor for medical history, physical exam, digital X-ray (with CAD4TB®) and AeoNose sampling. Participants will be offered voluntary HIV testing and counseling. In case of presumptive TB (estimated 20-30% of participants) two sputum samples will be taken, either spontaneous or saline-induced. One sample is tested with GeneXpert and the other with liquid mycobacterial culture. Cases of presumptive TB with both negative GeneXpert® and culture results will be followed-up after three and six months for repeat testing.

ELIGIBILITY:
Inclusion Criteria:

* All persons, either being a prisoner or employee, of the involved penal institutions after providing informed consent, including those with known active TB disease and/or currently on TB treatment

Exclusion Criteria:

* A potential participant who meets any of the following criteria will be excluded from participation in this study:

  1. Unable to exhale breath through the AeoNose™ during five minutes due to respiratory insufficiency
  2. Unable to stand in an upright position for the CXR
  3. Unable to communicate and comply with the instructions of the study team

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Volatile organic compound signal as measured with the AeoNose™ | Baseline/ change from baseline at 3 and 6 months
  The exhaled breath 'smell print' of each participant will be compared over time at baseline, 3 months and 6 months with sputum microbiology results and digital Chest Xray to establish sensitivity and specificity of electronic nose signal to diagnose Tuberculosis
Tuberculosis probablity score using Computed Automated detection software CAD4TB® on chest Xrays | Baseline/ change from baseline at 3 and 6 months
  Ranges from 0 to 100, where 0 would mean the lowest probability of having Tuberculosis and 100 would be the highest probability of having Tuberculosis.
Positive mycobacterial sputum test | Baseline/ change from baseline at 3 and 6 months
  positive GenXpert test and/or mycobacterial cultures are used to establish Tuberculosis diagnosis

SECONDARY OUTCOMES:
Comparison of predictive value of volatile organic compound signal with Tuberculosis Probability Score | Baseline/ change from baseline at 3 and 6 months
  comparison of correct positive predictions for active TB, with AeoNose (positive/ negative test result) and Cad4TB software from chest Xrays providing probability scores from 0-100 points
added value of the use of AeoNose and Cad4TB as a TB screening algorithm in vulnerable populations | Baseline/ change from baseline at 3 and 6 months
  evaluation of the combined use of both AeoNose and Cad4TB probability score to predict active TB

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Magis-Escurra, MD,PhD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Paraguay (2):
  - Buen Pastor, Asuncion, Central Department
  - UPI, Asuncion, Central Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: EUSAT-RCS TB research consortium — https://www.eusattb.net/

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT04407325/Prot_000.pdf
  • Informed Consent Form (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04407325/ICF_001.pdf